CLINICAL TRIAL: NCT01470274
Title: Safety of the CO-rebreathing Method in Stable Coronary Artery Disease and COPD Patients
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/1792
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Disease; Chronic Obstructive Pulmonary Disease
Keywords: Blood volume; CO-rebreathing; COPD; CVD
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to establish the safety of the CO-rebreathing method for measuring total blood and plasma volume in CAD patients. The working hypothesis is that the CO-rebreathing method is safe in use with coronary artery disease patients and that it does not cause myocardial ischemia or cardiovascular damage.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease
* Stable COPD
* Optimal medication

Exclusion Criteria:

* Unstable disease
* co-morbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable, optimally medicated coronary artery disease and COPD patients with LVEF ≥ 0.40 will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trine Karlsen, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Karlsen T, Leinan IM, Aamot IL, Dalen H, Stoylen A. Safety of the CO-Rebreathing Method in Patients with Coronary Artery Disease. Med Sci Sports Exerc. 2016 Jan;48(1):33-8. doi: 10.1249/MSS.0000000000000729. PMID 26672919